CLINICAL TRIAL: NCT05012709
Title: Developing a Healthy Care Environment in Psychiatry: A Study of Dose-response Relationship and the Evidence Based Multisensory Stimulation Intervention
Brief Title: A Study of Dose-response Relationship and the Evidence Based Multisensory Stimulation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jianan Psychiatric Center, Ministry of Health and Welfare (Other)
Collaborators: Taiwan Nurses Association (Other); National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Mei-Feng Lin, RN, Professor, Department of Nursing, College of Medicine, National Cheng Kung University, Jianan Psychiatric Center, Ministry of Health and Welfare
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JiananPsych
Record Dates: First submitted 2021-08-11; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Psychotic Disorders; Anxiety; Complementary Therapies; Clinical Trial
MeSH Terms: conditions — Psychotic Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: In total, 90 patients were randomly assigned to either the intervention or the control group. After a 2-week washout period, the intervention group was reassigned to the control and vice versa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group received six 30-minute MST sessions. During MST session, participants can choose their preferred sensory stimuli such as essential oil diffuses, music and so on.
  Interventions: Behavioral: multisensory stimulation therapy
- control group (No Intervention): The TAU group received usual routine care.

INTERVENTIONS:
Behavioral: multisensory stimulation therapy — The intervention group received six 30-minute MST sessions. During MST session, participants can choose their preferred sensory stimuli such as essential oil diffuses, music and so on.
  Arms: intervention group

SUMMARY:
Design: This parallel randomized controlled trial (RCT) was conducted according to the Consolidated Standards of Reporting Trials (CONSORT).

Methods: In total, 90 patients were randomly assigned to either the intervention or the control group. After a 2-week washout period, the intervention group was reassigned to the control and vice versa. The CONSORT checklist for RCT was reported. Psychotic symptoms, emotional reactions, behavioral relaxation responses and heart rates were assessed at 6 time points.

DETAILED DESCRIPTION:
This was a prospective randomized controlled trial with parallel groups following the Consolidated Standards of Reporting Trials and was approved by the Institutional Review Board of Jianan Mental Health Hospital (approval number Taiwan Nurses Association-1012023/ 12-002). Informed consent was obtained from all the subjects. Patients who had been hospitalized for schizophrenia, schizophreniform disorder, and schizoaffective disorder for more than 5 years according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (American Psychiatric Association, 2013) criteria were eligible to participate in the study. Patients who had a history of alcohol and drug abuse or could not concentrate on activities for at least 30 minutes were excluded from the study. As shown in the CONSORT diagram (Schulz et al., 2010), 109 patients were screened, 95 participants were enrolled by a research assistant and received interventions delivered by a nurse researcher. In the end, total 90 participants completely received multi-sensory stimulation therapy in a psychiatry institution in Southern Taiwan. None of the adverse events occurred. All patients were initially randomly assigned to either intervention or treatment as usual (TAU) group using a computer-generated random allocation sequence. The intervention group received six 30-minute MST sessions. During MST session, participants can choose their preferred sensory stimuli such as essential oil diffusers, music…etc.. The TAU group received usual routine care. After receiving either intervention or routine care, there was a 2-week washout period to clear the residual effects from the initial assigned group activities. Patients were then crossover into the other group where the process started over. Symptoms were assessed at baseline (T0), after the 1st session (T1), the 3rd session (T2) and the 6th session (T3). No important changes to the methods or trial outcomes were made after trial commencement.

Sample Size Calculation:

Sample size was calculated based on showing between group outcome differences after receiving MST according to a previous study (Cheng et al., 2017) of 60 patients who underwent the same comprehensive protocol. To achieve statistical significance p< 0.05, each parallel group of our study required at least 30 patients.

All the outcome assessments were by original assigned groups. Descriptive analysis was conducted for analyzing demographics and outcomes in all time points. Repeated Measurement of Analysis of Variance (ANOVA) was used to examine the effectiveness of MST between experimental and control groups. Effect size was determined using partial η2 that reflects the percentage of the variance in outcome variables explained by the independent variables.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients
* diagnosed with schizophrenia, schizophreniform disorder, and schizoaffective disorder for more than 5 years according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (American Psychiatric Association, 2013).
* aged above 20 years old

Exclusion Criteria:

* had a history of alcohol and drug abuse
* could not concentrate on activities for at least 30 minutes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-03-15 (Actual); Primary Completion 2013-01-10 (Actual); Study Completion 2013-03-10 (Actual)

PRIMARY OUTCOMES:
Change of Psychiatric Symptoms | Change from baseline BPRS at the sixth sessions (each session is 7 days).
  Brief Psychiatric Rating Scale (BPRS) consists of a series of 18 items that are used to assess the following psychotic symptoms: somatic concern, anxiety, emotional withdrawal, conceptual disorganization, guilt feelings, tension, mannerisms and posturing, grandiosity, depressive mood, hostility, suspiciousness, hallucinatory behavior, motor retardation, uncooperativeness, unusual thought content, blunted affect, excitement, and disorientation (Overall and Gorham, 1962). The total score range is between 0 (not present) and 18 (extremely severe). The reliability of BPRS in this study was acceptable (Cronbach's α = 0.71).
Change of Anxiety | Change from baseline HADS-A at the sixth sessions (each session is 7 days).
  The Hospital Anxiety and Depression Scale-Anxiety subscale (HADS-A) includes seven items. Each item is evaluated on a four-point (0 to 3) scale, with a total possible score range of 0 to 21. Scores of eight and higher indicate the possible presence of anxiety. The reliability of HADS-A in this study was acceptable (Cronbach's α = 0.67).
Change of Behavioral Relaxation | Change from baseline BRS at the sixth sessions (each session is 7 days).
  Behavioral Relaxation Scale (BRS) was administered to measure the motor elements of relaxation through observations of voluntary muscles by trained clinicians. Ten dimensions of postures were observed (e.g. breath, shoulders, hands… etc.) and behaviors were checked for indications of relaxation. The total score range of the BRS is between 0 (no relaxation) and 10 (relaxation).
Change of physiological responses | Change from baseline heart rate at the sixth sessions (each session is 7 days).
  Patients' Heart Rate, as an indicator of their responses to stress and tension, was measured by a wireless biofeedback system (MindMedia, Herten). The data was collected at a rate of 400 importing signals every minute.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Feng Lin, PhD, Study Chair — National Cheng Kung University
Locations (1):
- Mei-Feng, Lin, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Not shared with other research teams.

REFERENCES:
- [Background] American Psychiatric Association. (2013). Quick reference to the diagnostic criteria from DSM-V (p. 370). Washington, DC: APA.
- [Background] Overall, J. E., & Gorham, D. R. (1962). The brief psychiatric rating scale. Psychological reports, 10(3), 799-812. https://doi.org/10.2466%2Fpr0.1962.10.3.799
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Michultka DM, Poppen RL, Blanchard EB. Relaxation training as a treatment for chronic headaches in an individual having severe developmental disabilities. Biofeedback Self Regul. 1988 Sep;13(3):257-66. doi: 10.1007/BF00999174. PMID 3067751
- [Background] Cheng SC, Hsu WS, Shen SH, Hsu MC, Lin MF. Dose-Response Relationships of Multisensory Intervention on Hospitalized Patients With Chronic Schizophrenia. J Nurs Res. 2017 Feb;25(1):13-20. doi: 10.1097/jnr.0000000000000154. PMID 27310606
- [Background] Juszczak E, Altman DG, Hopewell S, Schulz K. Reporting of Multi-Arm Parallel-Group Randomized Trials: Extension of the CONSORT 2010 Statement. JAMA. 2019 Apr 23;321(16):1610-1620. doi: 10.1001/jama.2019.3087. PMID 31012939
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. Trials. 2010 Mar 24;11:32. doi: 10.1186/1745-6215-11-32. PMID 20334632